CLINICAL TRIAL: NCT04073966
Title: Magnetic Resonance Imaging Biomarkers for Radiation-Induced Neurocognitive Decline Following Stereotactic Radiosurgery of Newly Diagnosed Brain Metastases: An Observational Pilot Study
Brief Title: MRI Biomarkers for Radiation-Induced Neurocognitive Decline Following SRS of Newly Diagnosed Brain Mets
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1844
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; Neurocognitive Deficit; White Matter Alterations; Radiation Exposure
MeSH Terms: conditions — Brain Neoplasms; Leukoaraiosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain metastases are a source of much morbidity and mortality in adults with primary solid malignant tumors. With improvements in systemic therapy that prolong survival but have limited central nervous system penetration, patients with brain metastases are at increasing risk of developing and experiencing long-term side effects from treatment of brain metastases. The overarching goal of this study is to better understand the determinants of RT-associated changes in white and gray matter function and associated neurocognitive decline.

DETAILED DESCRIPTION:
The proposed study aims to provide novel and useful information for clinicians, both to help predict potential neurocognitive changes following SRS, and as a possible guide for SRS treatment alteration, whether through adjustment of dose or beam arrangements in relation to white matter tracts. In this observational pilot study of 20 patients, the association between RT-associated brain injury and neurocognitive function will be quantitatively assessed longitudinally over one year following SRS. The study team hypothesizes that, over this time, (1) there will be radiation dose-dependent reductions in regional white matter tract integrity and reduction in functional connectivity in the default mode network of gray matter, (2) there will be measurable decline in neurocognitive function, and (3) there will be an association between severity of radiation-induced brain injury on MRI and magnitude of neurocognitive functional decline. This association will relate, in part, to the location(s) affected.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of cancer
* Newly diagnosed brain metastasis being treated with SRS. Any extent of cranial disease permitted. Subsequent courses of SRS while on study permitted when clinically indicated.
* Patients are permitted to have undergone craniotomy and resection of metastasis/metastases if at least 1 other intact metastasis planned for definitive SRS is present. Receiving or previously received systemic therapy also permitted.
* Anticipated life expectancy at least 1 year
* Age ≥ 18 years
* Ability to read and comprehend written English and follow instructions in English
* Ability to provide informed consent

Exclusion Criteria:

* Previous radiation to the brain or head
* Previous malignancy - other than non-melanomatous skin cancer or cervical carcinoma in situ - and not disease-free for at least 3 years
* Previous severe head or brain injury
* History of a neurological disorder such as Epilepsy, Parkinson's, Alzheimer's, or Dementia
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed brain metastasis being treated with SRS.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Radiation-Induced White Matter Injury | One year after SRS completion
  Dose-dependent reductions in white matter integrity, as quantified by Diffusion Tensor MRI (DTI)-derived measures of change in diffusivity

SECONDARY OUTCOMES:
Changes in Functional Connectivity | One year after SRS completion
  Dose-dependent alterations in functional connectivity, especially for the subsystems of the Default Mode Network (DMN), as measured by resting state functional MRI
Neurocognitive Changes | One year after SRS completion
  Change in neurocognitive function, as measured by Delis-Kaplan testing, after SRS treatment

OTHER OUTCOMES:
Association between Changes in Functional Connectivity and Neurocognitive Changes | One year after SRS completion
  Correlation between magnitude of neurocognitive function decline and severity of radiation-induced brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Colette J Shen, MD, PhD, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology; Tong Zhu, PhD, DABR, Principal Investigator — University of North Carolina at Chapel Hill, Department of Radiation Oncology
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States